CLINICAL TRIAL: NCT04120428
Title: Effects of a 24-week Aquatic Exercise Training Program on Obstructive Sleep Apnea Severity in Elderly Women
Brief Title: Effects of Exercise on Obstructive Sleep Apnea Severity in Elderly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, Bruno Teixeira Barbosa, Master degree, Federal University of Paraíba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05768912401
Record Dates: First submitted 2019-10-07; First posted 2019-10-09 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Obstructive Sleep Apnea; Sleep-disordered Breathing; Sleep Disorder; Breathing-Related
Keywords: Aquatic exercise; Obstructive sleep apnea syndrome; Sleep
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Sleep Wake Disorders

STUDY DESIGN:
Intervention Model Description: Experimental group: 24-week aquatic exercise training program Control group: maintain life style routine as usual
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental protocol (Experimental): 24-week aquatic exercise training program
  Interventions: Other: Aquatic exercise training program
- Control protocol (No Intervention): Maintain lifestyle routine as usual

INTERVENTIONS:
Other: Aquatic exercise training program — The intervention will be performed in a pool in which the water surface line will remain in the imaginary line of the xiphoid process. Each season will last 50 minutes and will be divided in 3 phases as (1) warm-up (15 minutes), (2) main part (30 minutes) and (3) cool-down (5 minutes).
  Arms: Experimental protocol

SUMMARY:
Obstructive sleep apnea syndrome (OSAS) is defined as a total cessation of upper airway flow for at least 10 seconds. OSAS is considered under diagnosed and it is assessed by a full-night sleep polysomnography. Continuous positive airway pressure (CPAP) is considered the first line treatment to OSAS, however physical exercise has emerged as an adjunct and/or alternative strategy to CPAP in OSAS patients.

DETAILED DESCRIPTION:
Obstructive sleep apnea syndrome (OSAS), which comprises repeated episodes of total cessation of upper airway flow during sleep, is an underdiagnosed diasease and is closely related to major physiological desadjustments that compromises the systemic health of the human organism, including triggering death events; It is not surprising, therefore, that the prevalence of OSAS in adults and elderly varies widely.

Continuous positive airway pressure (CPAP) is the instrument used as first-line treatment for OSAS because it has significant responses in attenuating the severity of the syndrome, however, the design and logistical operation of the use of this instrument compromise the adherence to OSAS treatment .

In this sense, strategies such as regular exercise practice have promising initial results for the treatment of OSAS, despite the gaps that still exist due to the scarcity of studies completed in this area. To this end, it should be noted that studies evaluating the effects of exercise on the severity of OSAS deal mostly with adults / middle-aged adults in aerobic and / or resistance exercise practices performed in a terrestrial environment with alternation only of the ergometer used. Studies on physical exercise and OSAS in the elderly present marked scarcity and only one randomized clinical trial administered to elderly men was found.

The prescription of physical exercise for the elderly requires some precautions and precautions arising from the maladjustments that senescence promotes and that compromise the functionality of organic systems. These misfits include, among other things, the attenuation of lean mass with consequent reduction in muscle strength and dynamic balance; Such damages trigger, in the elderly, fall events that, linked to the reduction of bone mineral density due to aging, not infrequently lead to the physical and functional disability of the elderly.

Physical exercise performed in the aquatic environment, therefore, emerges as a safe and effective alternative in promoting physical and functional improvements for various populations due to the physical principles of water that promote buoyancy, reduction of joint stress, subjective perception of pain and exercise fatigue.

Therefore, the aim of the present study is to evaluate the effects of a 24-week aquatic training program on the severity of obstructive sleep apnea syndrome in older women and is justified in the emerging needs of 1) finding alternative solutions to CPAP use. , 2) use the practice of physical exercise as a tool in mitigating OSAS risk factors and severity; and 3) promote strategies of physical exertion as safe as they are effective for the elderly population to combat OSAS.

ELIGIBILITY:
Inclusion Criteria:

* Elderly women (60 years old or aged)
* Apparently healthy
* High risk to develop OSAS
* Diagnosed with moderate to severe OSAS
* No treated to OSAS with CPAP
* No use of any hypnotic medicine before or during the study

Exclusion Criteria:

* Cardiovascular, pulmonary or metabolic uncontrolled diseases
* Inability to perform the experimental protocol or keep the usual daily life
* Morbid obesity by body mass index

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Apnea-Hypopnea Index | Full-night sleep assessment: up to 8 hours
  Index which defines the OSAS severity. Is evaluated as events per hour by the polysomnography exam

SECONDARY OUTCOMES:
Self-related sleep quality | Face to face interview for 8 minutes
  Questionnaire score assessed by Pittsburgh Questionnaire, classifies self-related sleep quality as follows: as higher was the score as worse sleep quality is.
Daytime excessive somnolence | Face to face interview for 3 minutes
  Questionnaire score assessed by Epworth questionnaire which ranges from 0 to 18 and as higher was the score as higher the odds of the individual be considered with Daytime excessive somnolence.
Self-related quality of life | Face to face interview for 6 minutes
  Questionnaire score assessed by WHOQOL-Old questionnaire which ranges from 0 to 100 and as higher was the score as higher the odds of the individual be considered with good self-related quality of life.
Depressive symptoms | Face to face interview for 2 minutes
  Questionnaire score assessed by Geriatric Depressive Scale which ranges from 0 to 15 and as higher was the score as higher the odds of the individual be evaluated with depressive symptoms suspicious.
Oxygen consumption | Laboratory exam for 8-12 minutes
  This outcome will be assessed by a Cardiopulmonary exercise test in a cycle ergometer using Bruce Protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno T Barbosa, PhD Student, Principal Investigator — Federal University of Paraiba
Locations (1):
- Bruno Teixeira Barbosa, João Pessoa, Paraíba, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The authors will make the data available based on journal guidelines selected to make the article published.
Supporting Information: Study Protocol
Time Frame: The data will be available in the journal elected to publication as supplementary data.
Access Criteria: All the exercises which will be used in the 24-week aquatic exercise training program will be made available by making unknown the identity of the model.

REFERENCES:
- [Background] Bollens B, Reychler G. Efficacy of exercise as a treatment for Obstructive Sleep Apnea Syndrome: A systematic review. Complement Ther Med. 2018 Dec;41:208-214. doi: 10.1016/j.ctim.2018.10.002. Epub 2018 Oct 3. PMID 30477841
- [Background] Mendelson M, Bailly S, Marillier M, Flore P, Borel JC, Vivodtzev I, Doutreleau S, Verges S, Tamisier R, Pepin JL. Obstructive Sleep Apnea Syndrome, Objectively Measured Physical Activity and Exercise Training Interventions: A Systematic Review and Meta-Analysis. Front Neurol. 2018 Feb 22;9:73. doi: 10.3389/fneur.2018.00073. eCollection 2018. PMID 29520251
- [Background] Sengul YS, Ozalevli S, Oztura I, Itil O, Baklan B. The effect of exercise on obstructive sleep apnea: a randomized and controlled trial. Sleep Breath. 2011 Jan;15(1):49-56. doi: 10.1007/s11325-009-0311-1. Epub 2009 Nov 7. PMID 19898884
- [Background] Kline CE, Crowley EP, Ewing GB, Burch JB, Blair SN, Durstine JL, Davis JM, Youngstedt SD. The effect of exercise training on obstructive sleep apnea and sleep quality: a randomized controlled trial. Sleep. 2011 Dec 1;34(12):1631-40. doi: 10.5665/sleep.1422. PMID 22131599
- [Background] Barbosa BT, da Cruz Santos A, Frazao M, Petrucci TR, Cucato GG, Sarmento AO, Freitas EDS, de Lima AMJ, Brasileiro-Santos MDS. Obstructive sleep apnea does not impair cardiorespiratory responses to progressive exercise performed until exhaustion in hypertensive elderly. Sleep Breath. 2018 May;22(2):431-437. doi: 10.1007/s11325-017-1557-7. Epub 2017 Aug 24. PMID 28840546
- [Background] Tam S, Woodson BT, Rotenberg B. Outcome measurements in obstructive sleep apnea: beyond the apnea-hypopnea index. Laryngoscope. 2014 Jan;124(1):337-43. doi: 10.1002/lary.24275. Epub 2013 Jul 9. PMID 23794206